CLINICAL TRIAL: NCT05345899
Title: Evaluation of Plasma Vitamin C Levels in a Population of Chronic Rheumatism in Immuno-Rheumatology
Acronym: VitCRIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-PP-09
Record Dates: First submitted 2022-04-05; First posted 2022-04-26 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Lupus or SLE; Spondyloarthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic rheumatism (Other): Population of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain
  Interventions: Diagnostic Test: Evaluation of vitamin C level in plasma; Other: Evaluation of quality of life

INTERVENTIONS:
Diagnostic Test: Evaluation of vitamin C level in plasma — A protocol-specific blood test wil assess the vitamin C level in plasma
Other: Evaluation of quality of life — Several questionnaire will be completed by patients to evaluate quality of life: Analog and visual scale (EVA) pain, Neuropathic pain (DN) 4 questionnaire, EVA fatigue, Short Form (SF) 12 questionnaire and Hospital Anxiety and Depression scale (HAD questionnaire)

SUMMARY:
Scurvy is an almost forgotten carential pathology, caused by a deep vitamin C (or ascorbic acid) deficiency, a priori exceptional in industrialized countries. According to the French National Authority for Health standards, hypovitaminosis C is defined as a plasma vitamin C level of less than 23 μmol/L. This deficiency would affect 5 to 10% of the general population in industrialized countries and from 17% (clinical scurvy) to 47% (biological hypovitaminosis C) of vulnerable populations (malnutrition, hospitalized patients...). Vitamin C is essential for collagen synthesis. It plays a cofactor role in the synthesis of catecholamines precursors and takes action in synthesis of certain amino acids.

In rheumatology, pain is a recurring reason for consultation. In a context of treated chronic inflammatory rheumatism (RIC), while most of patients seem in remission or in reduced activity of their disease, all real-life studies show that 30 to 40% of them complain of residual pain, 70% of chronic fatigue and 20-25% of symptoms similar to secondary fibromyalgia. Currently, authors suggest the interest of vitamin C analgesic properties, especially in musculoskeletal pain, due to the role of ascorbic acid in neurotransmitters. Vitamin C would act as a cofactor for a family of biosynthetic and regulatory metalloenzymes. Thus, the authors suggest the potential of vitamin C in an analgesic mechanism involving the biosynthesis of opioid peptides.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years-old,
* followed for chronic inflammatory rheumatism (RIC): spondylo-arthritis (including spondylitis and psoriatic rheumatism) and lupus,
* with RIC in remission or low activity definec according to the following criteria: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) criteria and Bath Ankylosing Spondylitis Fonctional Index (BASFI) questionnaire for spondylitis and psoriatic rheumatism, Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) 2K score for lupus,
* having given written consent after written and oral information,
* member of the social security system,
* basic treatment for the disease not modified for at least 6 months, without modification at baseline
* persistence of painful complaints not objectively explained by his RIC.

Exclusion Criteria:

* pregnant or nursing patient,
* patient protected by law or under guardianship or curatorship, or not able to participate in a clinical trial under L.1121-16 article of French Public Health Regulations,
* patient participating in or having participated in another drug clinical trial in the month prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Describe prevalence of hypovitaminose C (ascorbemia below 23 µmol/L) in a population of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
  Among patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain and included in this study, the prevalence of hypovitaminosis C will be the proportion of patients with ascorbemia below 23 μmol/L measured at inclusion. Plasma ascorbemia will be measured using HPLC fluorimetric detection, using a Chromsystems kit.

SECONDARY OUTCOMES:
Age of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
Sexe of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
Socio-professional category of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
Type of disease of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
Length of illness of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
Type of disease's treatment for patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
Pain felt by patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
  Pain felt will be assessed with a visual and analog scale for pain which ranges from 0 (no pain) to 10 (maximum imaginable pain)
Tiredness felt by patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
  Tiredness felt will be assessed with a visual and analog scale for tiredness which ranges from 0 (no tiredness) to 10 (extreme tiredness).
Neuropatic pain felt by patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
  Neuropatic pain felt will be assessed with the neuropatic pain 4 (DN4) questionnaire, which ranges from 0 to 10. A score greater than 4 indicates a positive test.
Quality of life of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
  Quality of life will be assessed with the Short Form 12 (SF12) questionnaire.
Anxiety and depression of patients followed for chronic inflammatory rheumatism in remission or lupus in low activity, with chronic residual pain | at inclusion
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression (HAD) scale, splited in 2 scores which ranges from 0 to 21. A score less than 7 indicates a lack of symtomatology, a score between 8 and 10 indicates doubtful symptomatology and a score higher than 11 indicates a sure symptomatology.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No